CLINICAL TRIAL: NCT02231827
Title: A Study of the Balance Control During Gait : Comparison of Data Acquisition Between Force Plate and 3D Optoelectronic Gait Analysis System
Brief Title: Balance Control During Gait
Acronym: FREINAGE3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014/058/HP
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: subjects
MeSH Terms: interventions — Gait Analysis

ARMS (1):
- Gait analysis (Experimental)
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis — Subjects, barefoot and standing upright and motionless on a force plate, were instructed to walk for 10 m following a beep delivered by the experimenter. Two experimental conditions were tested: (i) the 'natural' gait condition where subjects walked normally and (ii) the 'fast' gait condition where subjects walked as fast as they could, taking large steps. Each subject performed 10 trials in each condition.
  Other Names: - Force plate; - 3D optoelectronic gait analysis system (VICON)

SUMMARY:
Gait and balance disorders are important public health problem necessitating studies to try to prevent falls. Many studies have dealt with spatiotemporal gait parameters or balance during quiet standing (posturography). Nevertheless, falls occurred predominantly during gait, and rarely during quiet standing. We have developed a tool to measure balance during gait : the braking of the center of mass (CM), a biomechanical parameter obtained from the vertical velocity of the CM recorded with a force plate.

In previous studies, we have shown that the braking of the CM was a physiological and a active mechanism, reflecting balance during gait. Unfortunately, the braking of the CM measured on a force plate provide an important intra-individual variability.

The 3D optoelectronic gait analysis system (VICON) also provide an estimation of the CM. The primary goal of this study is to compare intra-individual variability of the braking of the CM determined by a force plate or the 3D optoelectronic gait analysis system (VICON) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Between 20 and 40 years old
* Effective contraception for women of childbearing age

Exclusion Criteria:

* Neurological, vestibular, rheumatologic, orthopaedic disorders, which could influence gait and balance.
* Known spinal deformity
* Severe visual impairment : visual acuity less than 6/10
* Inability to stand and walk without assistance 15 meters
* Subjects without social security
* Subjects involved in another biomedical trial during this study
* Pregnant or breastfeeding women

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Braking of the center of mass index during gait initiation | 1 day
  Braking of the center of mass (CM), a biomechanical parameter obtained from the vertical velocity of the CM, determined by a force plate or a 3D optoelectronic gait analysis system (VICON).

SECONDARY OUTCOMES:
Braking of the center of mass index during locomotion | 1 day
  Braking of the center of mass (CM), a biomechanical parameter obtained from the vertical velocity of the CM, determined by a 3D optoelectronic gait analysis system (VICON).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie CHASTAN, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France